CLINICAL TRIAL: NCT05297409
Title: Hyperkalemia Registry An Observational Prospective Cohort Study for Long-term Management of Hyperkalemia in Patients With Chronic Kidney Disease or Heart Failure
Brief Title: An Observational Prospective Cohort Study for Long-term Management of Hyperkalemia in Patients With Chronic Kidney Disease or Heart Failure
Acronym: HK registry
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D9480R00027
Record Dates: First submitted 2022-03-17; First posted 2022-03-28 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-07

CONDITIONS: Hyperkalemia
MeSH Terms: conditions — Hyperkalemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Hyperkalemia patient with Chronic kidney disease
- hyperkalemia patient with heart failure

SUMMARY:
This prospective observational research will be conducted to assess the burden of hyperkalemia including treatment and disease burden of patients in a long-term continuous care from various aspects including adherence to the medication for hyperkalemia and HR-QoLs.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hyperkalemia who meet the following criteria:

  1) Being treated with potassium binders for hyperkalemia at the time of enrolment, and having started receiving potassium binders within 6 months before enrolment
* Having been diagnosed as CKD (≥stage 3b) or HF diagnosed by investigators, and as defined below:

  1) CKD is diagnosed based on the CKD guidelines issued by the Japanese Society of Nephrologyxxix as being either or both of condition 1 and 2 for ≥3 months

  1-i) Clear signs of kidney impairment based on the results of urinalysis, imaging, blood test, or biopsy. Presence of proteinuria, especially more than 0.15 g/gCr (albuminuria more than 30 mg/gCr).

  1-ii) GFR <45 mL/min/1.73m2

  2) Patients with HFwill be enrolled if patients meet following criteria: 2-i) NYHA class II-IV, within 6 months 2-ii) Patients with a diagnosis or history of heart failure, hospitalization, and laboratory records of any of the following; NT-proBNP≥400 pg/ml or BNP≥100 pg/ml, or pathological findings such as abnormal cardiac function by UCG/CT/MRI/catheterization/nuclear medicine examination
* Provision of signed, written, and detailed informed consent

Exclusion Criteria:

* Currently on any chronic RRT (including hemodialysis or peritoneal dialysis >30 days, or kidney transplant) within 6 months before enrolment
* Patients with acute kidney injury (AKI)* within 6 months before enrolment
* Patients with acute heart failure within 3 months before enrolment
* Patients who received blood transfusion within 6 months before enrolment
* Patients with active malignancy or whose life expectancy is less than 6 months
* GI disturbance, chronic diarrhoea, or GI stoma if, as judged by the investigators, that condition or its treatment has an important impact on S-K values
* Autoimmune disease if, as judged by the investigators, that condition or its treatment has an important impact on S-K values
* Patients who are suspected, on the basis of laboratory data, to have pseudohyperkalemia (abnormality in the sample, a history of severe leukocytopenia or thrombocytopenia)
* Patients with recent traumatic injury
* Patients who are pregnant, lactating, or planning to become pregnant
* Current participation in a clinical trials, i.e. an interventional studies
* Presence of a condition that, in the opinion of the investigator, i) would places the subject at undue risk, or ii) would potentially jeopardizes the quality of the data to be generated, or iii) would prevent the patient from performing protocol-defined tasks for physical or mental reasons, or iv) would prevent the patient from understanding the contents of the self-administered questionnaire and responding to its questions on his/her own, or v) would, for some other reason, make the patient inappropriate for this study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult out-patients with CKD stage 3b, stage 4, or stage 5, or with HF (NYHA class II-IV) who are being treated with potassium binders for hyperkalemia at the time of enrolment, and who started receiving potassium binders within 6 months before enrolment
Sampling Method: Non-Probability Sample
Enrollment: 352 (Actual)
Dates: Start 2022-05-21 (Actual); Primary Completion 2024-08-28 (Actual); Study Completion 2024-08-28 (Actual)

PRIMARY OUTCOMES:
Patient characteristics including socio-demographic variables, severity of disease and comorbidities | 6 month
Health-Related Quality of Life | 6 month
Serum Potassium | 6 month

SECONDARY OUTCOMES:
Nutritional status | 6 month
Status of metabolic acidosis | 6 month
Use of healthcare resource | 6 month

OTHER OUTCOMES:
Onset or worsening of HF, any rapid decline in kidney function, GI symptoms and peripheral edema | 6 month

CONTACTS AND LOCATIONS:
Locations (28):
- Japan (28):
  - Research Site, Kasugai, Aichi-ken
  - Research Site, Nagaoka, Aichi-ken
  - Research Site, Matsudo, Chiba
  - Research Site, Chikushino-shi, Fukuoka
  - Research Site, Iizuka-shi, Fukuoka
  - Research Site, Kitakyushu-shi, Fukuoka
  - Research Site, Takasaki, Gunma
  - Research Site, Fukuyama, Hiroshima
  - Research Site, Hirosima-shi,Naka-ku, Hiroshima
  - Research Site, Hakusan, Ishikawa-ken
  - Research Site, Kanazawa, Ishikawa-ken
  - Research Site, Kawasaki-shi,Kawasaki-ku, Kanagawa
  - Research Site, Kawasaki-shi,Miyamae-ku, Kanagawa
  - Research Site, Kuwana, Mie-ken
  - Research Site, Sendai, Miyagi
  - Research Site, Azumino, Nagano
  - Research Site, Ueda, Nagano
  - Research Site, Nagaoka, Niigata
  - Research Site, Osaka-shi,Kita-ku, Osaka
  - Research Site, Sakai, Osaka
  - Research Site, Bunkyo, Tokyo
  - Research Site, tabashi City, Tokyo
  - Research Site, Kagoshima
  - Research Site, Kochi
  - Research Site, Shizuoka
  - Research Site, Tochigi
  - Research Site, Toyama
  - Research Site, Yamagata

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Shibagaki Y, Yamazaki H, Wakita T, Ware JE, Wang J, Onishi Y, Yajima T, Sada KE, Yamamoto Y, Fukuhara S. Impact of treatment of hyperkalaemia on quality of life: design of a prospective observational cohort study of long-term management of hyperkalaemia in patients with chronic kidney disease or chronic heart failure in Japan. BMJ Open. 2023 Dec 14;13(12):e074090. doi: 10.1136/bmjopen-2023-074090. PMID 38101840
- See also: D9480R00027_Redacted_CSR_synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9480R00027&attachmentIdentifier=49ab409f-d5fa-4272-82f4-6783e5fef039&fileName=D9480R00027_Redacted_CSR_synopsis.pdf&versionIdentifier=